CLINICAL TRIAL: NCT02676531
Title: Effects of Walking Meditation on Vascular Function in Breast Cancer Patients Receiving Anthracyclines Chemotherapy
Brief Title: Walking Meditation Exercise in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr.Daroonwan Suksom, Faculty of sports science, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SPSC-5
Record Dates: First submitted 2016-01-17; First posted 2016-02-08 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Walking Meditation; Vascular Function; Flow-mediated dilatation; Breast Cancer Patients; Anthracyclines Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Walking Meditation (Experimental): Walking Meditation program will be based on aerobic walking exercise combined with Buddhist meditation. The subjects will perform walking while listening to the sound "Budd" and "Dha" and squeeze rubber balls according to the sound in order to practice mindfulness while walking. In phase 1 (week 1-6), Walking Meditation will be conducted at initial moderate intensity (41-50% heart rate reserve) 3 sets, 10 minutes per set and rest 3 minutes between set In phase 2 (week 7-12), the training intensity will be increased to ultimate moderate intensity (51-60% heart rate reserve) 3 sets, 15 minutes per set and rest 3 minutes between set. In both phases of the training, the frequency of Walking Meditation training is three times a week.
  Interventions: Other: Exercise
- No Walking meditation (No Intervention): keep regular activities, sedentary life style.

INTERVENTIONS:
Other: Exercise — Walking meditation exercise program
  Arms: Walking Meditation

SUMMARY:
This study is to evaluate the effects of Walking Meditation on vascular function in breast cancer patients receiving Anthracyclines chemotherapy

DETAILED DESCRIPTION:
Walking Meditation program will be based on aerobic walking exercise combined with Buddhist meditation. The subjects will perform walking while listening to the sound "Budd" and "Dha" and squeeze rubber balls according to the sound in order to practice mindfulness while walking. In phase 1 (week 1-6), Walking Meditation will be conducted at initial moderate intensity (41-50% heart rate reserve) 3 sets, 10 minutes per set and rest 3 minutes between set In phase 2 (week 7-12), the training intensity will be increased to ultimate moderate intensity (51-60% heart rate reserve) 3 sets, 15 minutes per set and rest 3 minutes between set. In both phases of the training, the frequency of Walking Meditation training is three times a week.

ELIGIBILITY:
Inclusion Criteria:

1. The inclusion criteria included stage 1-2 of Breast cancer patients after an operation with or without Hormone Receptor Positive and HER2 Positive.
2. All participants will be planned to use Anthracyclines chemotherapy in next 1 month by oncologist.
3. All participants did not participate in any exercise training in the past 6 months
4. All participants are free from acute or chronic renal failure, Heart Failure, Myasthenia gravis, pregnancy and history of smoke.

Exclusion Criteria:

1. Participants will be excluded if they dropped out or completed less than 80% of the training schedule.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vascular reactivity | baseline, up to 12 weeks
  Vascular reactivity or brachial artery flow-mediated dilatation (FMD) will be assessed with the ultrasound equipment (CX50, Philips, USA), using the blood occlusion technique on the forearm. The brachial artery will be illustrated above the antecubital fossa in the longitudinal plane. Brachial FMD will be measured at resting and the cuff placed around the forearm will be inflated to 50 mmHg above systolic blood pressure for 5 minutes and then deflated for 5 minutes of recovery. FMD will be calculated from the formula FMD= (D2-D1) x100/D1 when D1 is the brachial artery diameter at baseline, D2 is the maximal post-occlusion brachial artery diameter.

SECONDARY OUTCOMES:
Change from baseline in Intima-Media Thickness: IMT | baseline, up to 12 weeks
  Intima-Media Thickness will be assessed with the ultrasound equipment (CX50, Philips, USA).
Change from baseline in Peripheral arterial stiffness | baseline, up to 12 weeks
  Pulse wave velocity (brachial-ankle PWV) measurement will be assessed by using Omron Colin VP1000.
Change from baseline in venous blood flow | baseline, up to 12 weeks
  Venous blood flow will be assessed with the ultrasound equipment (CX50, Philips, USA). The Basilic vain will be illustrated in the longitudinal plane. Venous blood flow will be measured at resting and squeezing hand for 3 minutes and 5 minutes of recovery. Venous blood flow will be calculated from the formula CSA x V when CSA is the cross sectional area of Basilic vain, V is the velocity in vessel.
Change from baseline in blood chemistry | baseline, up to 12 weeks
  1. Nitric oxide (NO) will be measured in serum samples with the commercial assay kit.
  2. Malondialdehyde (MDA) will be determined in plasma samples using the High Performance Liquid Chromatography (HPLC).
  3. Interleukin-6 (IL-6) will be measured in serum samples with the ELISA kit.
  4. hs-CRP will be measured in serum samples with the ELISA kit.
Change from baseline in Maximal oxygen consumption | baseline, up to 12 weeks
  Maximal oxygen consumption (VO2max) will be assessed by Bruce Ramp Protocol for treadmill test with Stationary Gas Analyzer (Vmax™ Encore 29 system, Yorba Linda, CA).
Change from baseline in Cardiac output and stroke volume | baseline, up to 12 weeks
  Cardiac output and stroke volume will be measured by using Physioflow (PF07 enduro).
Change from baseline in Body Mass Index (BMI) | baseline, up to 12 weeks
  Body Mass Index (BMI) will be measured using Body Composition Analyzer (Model ioi 353, Jawon Medical Co. Ltd., Korea). BMI will be calculated by dividing weight in kilograms by height in metres squared.
  Unit of BMI is kg/m2.
Change from baseline in stress indicators | baseline, up to 12 weeks
  Serum cortisol will be measured with cortisol kit.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siripanya S, Parinyanitikul N, Tanaka H, Suksom D. Home-Based Buddhist Walking Meditation Mitigates Cardiotoxicity of Anthracycline Chemotherapy in Breast Cancer Patients: A Randomized Controlled Trial. J Integr Complement Med. 2023 Sep;29(9):562-573. doi: 10.1089/jicm.2022.0778. Epub 2023 Apr 10. PMID 37036793